CLINICAL TRIAL: NCT04362306
Title: Radiation Oncology Patient Medical Physics Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CTMS# 19-0182
Record Dates: First submitted 2020-04-14; First posted 2020-04-24 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Anxiety; Patient Satisfaction; Radiation Therapy
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Planned Intervention (Experimental): Patients will be scheduled for CT (computed tomography ) simulation for radiation treatment planning. Prior to simulation, patients will be asked to complete anxiety and patient satisfaction questionnaires. Following completion of the questionnaires, each patient will receive the first intervention with a member of the medical physics team to review the process of simulation, treatment planning, and subsequent treatment. This meeting will last approximately 15 minutes and at this time, the team member will explain that they are the primary resource for all the technical aspects related to the patient's treatment. Additionally, they will identify and address any concerns that patients or their caregivers have with radiation treatment and the patient will be shown the simulation infographic. The patient will then be asked to complete a second set of anxiety and patient satisfaction questionnaires and will then undergo the planned simulation.
  Interventions: Behavioral: Planned Intervention
- No Planned Intervention (Active Comparator): After patients are enrolled into this study, they will be scheduled for CT simulation for radiation treatment planning. Prior to simulation, patients will receive anxiety and patient satisfaction questionnaires to complete
  Interventions: Behavioral: No planned intervention

INTERVENTIONS:
Behavioral: Planned Intervention — Intervention with a member of the medical physics team to review the process of simulation, treatment planning, and subsequent treatment. This meeting will last approximately 15 minutes and at this time, the team member will explain that they are the primary resource for all the technical aspects related to the patient's treatment. Additionally, they will identify and address any concerns that patients or their caregivers have with radiation treatment and the patient will be shown the simulation infographic.
  Arms: Planned Intervention
Behavioral: No planned intervention — Anxiety and patient satisfaction questionnaires will be completed prior to CT simulation.
  Other Names: Control group
  Arms: No Planned Intervention

SUMMARY:
This investigation is designed to be a two-arm, non-randomized prospective phase 2 study evaluating the impact of medical physicist patient intervention on the anxiety level and patient satisfaction of patients undergoing a course of radiation therapy. The goal is to demonstrate that these interventions will have a significantly positive impact on the overall well-being of the oncology patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Patients receiving treatment in the outpatient setting.
* Patients with an Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0, 1, or 2.

Exclusion Criteria:

* Patients receiving a single fraction of treatment.
* History of Prior Radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Anxiety Inventory | Baseline to last treatment (up to 9 weeks)
  The change in score from 6 questions in the validated short-form of the Spielberger State-Trait Anxiety Inventory (STAI).10 The mean medical physics intervention cohort anxiety score will be calculated at each of the 4 time points and compare to the same time points for the control cohort.
Patient Satisfaction | Baseline to last treatment (up to 9 weeks)
  Change in mean Function Assessment of Chronic Illness Therapy Treatment Satisfaction Patient Satisfaction score for the control and intervention groups will be compared.

SECONDARY OUTCOMES:
Medical competency/health literacy of Spanish speaking patients | Prior to CT simulation
  Analyze medical competency/health literacy through a one-time, 3-question medical competency questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wagner, MD, MBA, Principal Investigator — University of Texas
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No